CLINICAL TRIAL: NCT05845996
Title: A Randomized, Double-blind, Parallel Design, Placebo-controlled Single and Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous and Subcutaneous Doses of SAR441344 in Healthy Adult Subjects
Brief Title: Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous and Subcutaneous Single and Repeated Doses of SAR441344 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDU15525-TDR15526; U1111-1217-2909 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — keyhole-limpet hemocyanin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR441344 (Experimental): Single or multiple Ascending dose of SAR441344 Dose 1 administered intravenously and/or subcutaneously
  Interventions: Drug: SAR441344; Biological: Keyhole limpet hemocyanin
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: placebo; Biological: Keyhole limpet hemocyanin

INTERVENTIONS:
Drug: SAR441344 — Solution for intravenous/subcutaneous injection
  Arms: SAR441344
Drug: placebo — Solution for intravenous/subcutaneous injection
  Arms: placebo
Biological: Keyhole limpet hemocyanin — Subcutaneous Lyophilized powder for reconstitution

SUMMARY:
Primary Objective is the tolerability and safety of ascending single and repeated intravenous infusion (IV) and/or subcutaneous (SC) administration of SAR441344

DETAILED DESCRIPTION:
The study duration of Part 1 is approximately 22 weeks, including a treatment period of 1 day; The study duration of Part 2 is approximately 26 weeks for each subject, including a treatment period of 29 days.

ELIGIBILITY:
Inclusion criteria

- Having given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria

- Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with adverse event(AE) | From baseline to day 127
  Number of participants with AE from baseline to day 127
Part 2: Number of participants with adverse event (AE) | From baseline to day 155
  Number of participants with AE from baseline to day 155

SECONDARY OUTCOMES:
Assessment of PK parameter: Cmax | From Day 1 to Day 127 and to Day 155
  Maximum plasma concentration (Cmax) observed
Assessment of PK parameter: tmax | From Day 1 to Day 127 and Day 155
  First time to reach Cmax (tmax)
Assessment of PK parameter: AUClast | From Day 1 to Day 127
  Area under the plasma concentration versus time curve from time zero to the real time
Assessment of PK parameter: AUC | Area under the plasma concentration versus time curve extrapolated to infinity
  From Day 1 to Day 127
Assessment of PK parameter: AUC0-tau | From day 1 to Day 155
  Area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (336 hours)
Assessment of PK parameter: Ctrough | From Day 1 to Day 155
  Plasma concentration observed just before treatment administration during repeated dosing
Assessment of PK parameter: t1/2z | From Day 1 to Day 127 and Day 155
  Terminal half-life associated with the terminal slope (λz)
Assessment of PK parameter: CL(/F) | Apparent total body clearance of a drug from the plasma
  From Day 1 to Day 127
Assessment of PK parameter: CLss(/F) | Apparent total body clearance of a drug from the plasma
  From day 1 to Day 155
Anti-SAR441344 antibodies | From Day 1 to Day 127 and Day 155
  Number of subjects with treatment emergent anti-drug antibody formation
Assessment of anti-KLH IgG and IgM | From Day 1 to Day 127 and Day 155
  Measurement of anti-KLH IgG and IgM levels in response to KLH immunization
AE attributed to KLH immunization | From Day 1 to Day 127 and Day 155
  Number of participants with AE attributed to KLH immunization

CONTACTS AND LOCATIONS:
Locations (1):
- PPD-Site Number:8400001, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TDU15525 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25457&tenant=MT_SNY_9011
- See also: TDR15526 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25444&tenant=MT_SNY_9011